CLINICAL TRIAL: NCT03071874
Title: A Single Arm Phase II Study Of The Dual mTORC1/mTORC2 Inhibitor Vistusertib (AZD2014) Provided On An Intermittent Schedule For Sporadic Patients With Grade II-III Meningiomas That Recur Or Progress After Surgery And Radiation
Brief Title: Vistusertib (AZD2014) For Recurrent Grade II-III Meningiomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Scott R. Plotkin, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-563; R01CA201130-01A1 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-03-07 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Meningioma
Keywords: Meningioma
MeSH Terms: conditions — Meningioma | interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD2014 (Experimental): * AZD2014 will be administered orally at a pre-determine dose
  * Twice daily for two consecutive days out of every seven days
  * Cycles will last 28 days
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014 — AZD2014 is a dual mTORC1/mTORC2 inhibitor
  Other Names: vistusertib

SUMMARY:
This research study is studying a chemotherapy as a possible treatment for Meningiomas (recurrent).

The study intervention involved in this study is:

--AZD2014 (vistusertib)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved AZD2014 as a treatment for any disease.

The goal of this clinical research study is to learn if the study drug AZD2014 can shrink or slow the growth of meningioma. Based on laboratory research, the cellular pathways which are blocked by AZD2014 are important for the growth and survival of meningiomas. Further, treatment of meningioma cells in the laboratory has resulted in decreased survival of tumor cells. As such, the purpose of this research is to see whether treating recurrent grade 2-3 meningioma with AZD2014 will result in tumor size stabilization or shrinkage. The safety of AZD2014 will also be studied. The physical state, the symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if AZD2014 is safe and effective in participants with this condition.

AZD2014 is being studied in patients with various cancers as a single agent (a drug that is used alone to treat the cancer) or in combination with a number of well known anticancer therapies. Previous studies have also allowed investigators to determine the best dose and frequency of AZD2014 to achieve anti-tumor effects while reducing the likelihood of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed intracranial meningioma, grade II-III,that has recurred or progressed at previous treatment.
* Participants must be willing and able to undergo regular MRI scans of the brain.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm with MRI, performed within 30 days prior to study registration.
* Patients must have received prior surgical resection and radiation therapy for the progressive meningioma.
* Patients must have received less than three prior chemotherapy regimens for progressive meningioma.
* Patients must have available an archival paraffin tumor block sufficient to generate at least 20 unstained slides; or, if a paraffin tumor block is unavailable, at least 20 unstained slides.
* Age ≥ 18 years at the time of study enrollment.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A) with no deterioration over the previous 2 weeks.
* Life expectancy of greater than three months
* Within 14 days of study registration, participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * hemoglobin ≥90 g/L
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 x institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Serum creatinine ≤1.5 x institutional upper limit of normal concurrent with creatinine clearance ≥50 mL/min (measured or calculated by Cockcroft and Gault equation), confirmation of creatinine clearance is only required when creatinine is >1.5xULN
  * Urine protein ≤1+ on urine dipstick (if 2+ seen on first test, re-test at least 24 hours later)
  * PT/INR/PTT (aPTT) <1.5x institutional upper limit of normal
* The effects of AZD2014 on the developing human fetus are unknown. For this reason and because mTOR kinase inhibiting agents are known to be teratogenic, female patients must be willing to use 2 forms of highly effective contraception (per institution standards) from the time of screening until four weeks after discontinuing study, must not be breast feeding, and must have a negative pregnancy test prior to start of dosing if of child bearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening: (1) post-menopausal women, defined as either women aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments, or (2) women under 50 years old who have been amenorrheic for at least 12 months following the cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels in the postmenopausal range for the institution. Alternatively, women must have documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

Male patients should either be surgically sterile or willing to use an effective barrier method of contraception during the study and for 16 weeks following the last dose of study treatment if sexually active with a female of childbearing potential. If not done previously, storage of sperm prior to receiving AZD2014 will be advised to male patients with a desire to have children.

* Ability to understand and the willingness to sign a written informed consent document prior to any study specific procedures, sampling, and analyses.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* Participants with a clinical diagnosis of NF2 (either by NIH or Manchester criteria) or with a molecular diagnosis of NF2
* Participants who received biopsy only or have received more than 2 prior courses of radiation for meningioma
* Participants who have had chemotherapy, radiotherapy, biological therapy, immunotherapy or other anticancer agents within 14 days (six weeks for nitrosoureas or mitomycin C) prior to entering the study.
* With the exception of alopecia, any unresolved toxicities from prior anti-tumor treatments (excluding corticosteroids) should be no greater than CTCAE (Version 4.0) Grade 1 at the time of study entry.
* Major surgery within four weeks prior to entry to the study (excluding placement of vascular access), or minor surgery (excluding tumor biopsies) within 14 days of first dose of study treatment.
* Participation in another clinical study with an investigational product during the last 21 days.
* History of hypersensitivity to active or inactive excipients of AZD2014 or drugs with a similar chemical structure or class to AZD2014.
* Exposure to strong or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) and BCRP if taken within the stated washout periods before the first dose of study treatment (see Appendix B)
* Exposure to specific substrates of the drug transporters OATP1B1, OATP1B3, MATE1 and MATE2K within the appropriate wash-out period (a minimum of 5 x reported elimination half-life) before the first dose of study treatment (see Appendix B)
* Any hematopoietic growth factors (e.g., filgrastim [granulocyte colony-stimulating factor; G-CSF], sargramostim [granulocyte-macrophage colony-stimulating factor; GM-CSF]) within 14 days prior to receiving study treatment.
* Pre-treatment with other mTOR inhibitors may be allowed and should be discussed with the medical monitor.
* Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Previous meningioma progression during treatment with other mTORC1/2 inhibitors (but not mTORC1 inhibitors such as everolimus or other rapalogs).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, severe hepatic impairment, interstitial lung disease (bilateral, diffuse, parenchymal lung disease), uncontrolled chronic renal diseases (glomerulonephritis, nephrotic syndrome, Fanconi Syndrome or renal tubular acidosis), current unstable or uncompensated respiratory or cardiac conditions, uncontrolled hypertension, active bleeding diatheses, active hepatitis B or C infection, known active human immunodeficiency virus (HIV) infection, or psychiatric illness/social situations that would limit compliance with study requirements. Screening for chronic conditions is not required.
* History of other malignancies, except: Malignancy treated with curative intent and with no known active disease present for ≥5 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician, (2) adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, (3) adequately treated carcinoma in situ without evidence of disease, or (4) Gleason 6 prostate cancer under observation.
* Patients who have experienced any of the following procedures or conditions currently or in the preceding 12 months:

  * coronary artery bypass graft
  * angioplasty
  * vascular stent
  * myocardial infarction
  * angina pectoris
  * congestive heart failure New York Heart Association Grade ≥2 (ventricular arrhythmias requiring continuous therapy)
  * supraventricular arrhythmias including atrial fibrillation, which are uncontrolled
  * hemorrhagic or thrombotic stroke, including transient ischemic attacks or any other central nervous system bleeding
  * History of drug abuse or alcohol abuse, as judged by the Investigator
* Abnormal echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) at baseline (left ventricular ejection fraction [LVEF] <55%). Appropriate correction to be used if a MUGA is performed.
* Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis.
* Mean resting corrected QT interval (QTc), calculated using Fridericia's formula, > 470 msec obtained from 3 electrocardiograms (ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes within 12 months of the patient entering in the study.
* Patients with uncontrolled Type II (HbA1c >8% assessed locally) as judged by the investigator or abnormal fasting glucose value defined as >126 mg/dL (>7 mmol/L).
* Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age). See appendix B for a list of medications.
* Vaccinated with live, attenuated vaccines within four weeks of the first dose of study drug.
* Judgment by the Investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
* Pregnant women are excluded from this study because AZD2014 is an mTORC1/2 inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD2014, breastfeeding should be discontinued if the mother is treated with AZD2014.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2014. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca, CRO staff, and/or staff at the CPU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 months
  proportion of patients alive and without progression

SECONDARY OUTCOMES:
Overall Survival | 2 years
  time from registration to death due to any cause, or censored at date last known alive
Radiographic Response Rate | 2 years
  proportion of patients with complete or partial radiographic response
Duration of Radiographic Response | 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Frequency of Adverse Events | 2 years
  frequency of subjects experiencing a specific adverse event will be tabulated grade, and relationship to study drug

CONTACTS AND LOCATIONS:
Overall Officials: Scott R. Plotkin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Massachusetts general Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No